CLINICAL TRIAL: NCT06581627
Title: A Single-centre, Open-label, Single-group Study Investigating the Pharmacokinetics, Safety and Tolerability After a Single Dose of Oral Etavopivat in Healthy Chinese Participants
Brief Title: A Research Study Looking at a Single Dose of Etavopivat in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7535-7704; U1111-1294-7463 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers; Sickle Cell Disease; Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Etavopivat (Experimental): Participants will be administered a single dose of 2 tablets of etavopivat together.
  Interventions: Drug: Etavopivat

INTERVENTIONS:
Drug: Etavopivat — 2 tablets of Etavopivat will be administered in fasted state via oral route

SUMMARY:
The study tests a new medicine called etavopivat in healthy Chinese participants. During the study, the participant will be given 1 dose of the study medicine. A dose is 2 tablets which are swallowed together with a cup of water. The study doctor will measure how much of the study medicine is in the blood as time passes. After the dose is given, the study will last for 7 to 9 days. The participants will attend a screening visit 2 to 28 days before they are given the study medicine. The participant will have 6 clinic visits in total. As part of the study, participant will stay overnight at the clinic for 3 nights. In some cases the doctor may decide that participant need to stay more nights. Participant will have blood tests and other health assessments at all 6 visits. Women cannot take part if pregnant, breast-feeding or plan to get pregnant during the study period. If the participant do take part in the study, participant will need to refrain from certain activities and behaviours for up to 3 months before taking the study medicine. Participant will also need to go without food and drinks other than water in the 10 hours before and 4 hours after taking the medicine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Chinese participants.
* Age 18-45 years (both inclusive) at the time of signing the informed consent form.
* Body mass index (BMI) between 18.0 and 33.0 kg/m^2 (both inclusive) at screening.
* Body weight greater than or equal to 40.0 kg at screening.
* Considered to be generally healthy based on the medical history, physical examination and the results of vital signs, electrocardiogram (ECG) and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive methods.
* Participation (i.e., signed informed consent) in any other interventional clinical study within 90 days or 5 times the half-life of the previous investigational medical product (IMP) (if known), whichever is longer before screening.
* Any disorder, unwillingness or inability, which in the investigator's opinion might jeopardise the participant's safety or compliance with the protocol.
* Use of any medication with unknown or unspecified content within 90 days before screening.
* Use of prescription medicinal products or non-prescription drugs (including Chinese traditional medicine or local medicine) within 14 days before screening, as declared by the participant, apart from:
* Acceptable contraceptive methods
* Hormone replacement therapy (for menopausal females)
* Over-the-counter topical medications known to not reach systemic circulation
* Occasional use of:
* Acetaminophen up to 2 grams (g) (4 x 0.5 g) daily
* Ibuprofen up to 2.4 g (4 x 0.6 g) daily
* Acetylsalicylic acid up to 2.4 g (4 x 0.6 g) daily
* Is unable to refrain from or anticipates the use of any drug known to be a strong or moderate inhibitor or inducer of uridine 5'-diphospho glucuronosyltransferase (UGT) enzymes, cytochrome P450 (CYP) 3A4, CYP2C9 or permeability glycoproteins (P-gp), including St. John's Wort, for 28 days prior to dosing and throughout the study
* Is unable to refrain from or anticipates the use of any medications or substances prohibited in the study
* Use of tobacco and nicotine products, defined as any of the following:
* Has used any product containing tobacco or nicotine within 90 days prior to screening
* Not willing to refrain from the use of any product containing tobacco or nicotine throughout the study
* Positive nicotine test at screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
AUC0-inf,etavopivat: Area under the etavopivat plasma concentration-time curve from 0 hours and extrapolated to infinity after a single dose | From 0 to 120 hours after investigational medicinal product (IMP) administration (day 6)
  Measured in hour*nanogram/millilitre (h*ng/mL).
Cmax,etavopivat: Maximum observed etavopivat plasma concentration after a single dose | From 0 to 120 hours after investigational medicinal product (IMP) administration (day 6)
  Measured in nanograms/millilitre (ng/mL).
Weight-adjusted AUC0-inf,etavopivat: Area under the etavopivat plasma concentration-time curve from 0 hours and extrapolated to infinity after a single dose divided by body weight | From 0 to 120 hours after investigational medicinal product (IMP) administration (day 6)
  Measured in(hour*nanogram/millilitre)/kilograms ((h*ng/mL)/kg).
Weight-adjusted Cmax,etavopivat: Maximum observed etavopivat plasma concentration after a single dose divided by body weight | From 0 to 120 hours after investigational medicinal product (IMP) administration (day 6)
  Measured in (nanograms/millilitre )/kilogram ((ng/mL)/kg).
AUC0-last,etavopivat: Area under the etavopivat plasma concentration-time curve from0 hours to the time of last quantifiable concentration | From 0 to 120 hours after investigational medicinal product (IMP) administration (day 6)
  Measured in hour*nanogram/millilitre (h*ng/mL).
tmax,etavopivat: Time to maximum observed etavopivat plasma concentration after a single dose | From 0 to 120 hours after investigational medicinal product (IMP) administration (day 6)
  Measured in hour (h).
t½,etavopivat: Terminal half-life for etavopivat after a single dose | From 0 to 120 hours after investigational medicinal product (IMP) administration (day 6)
  Measured in hour (h).
CL/F etavopivat: Apparent plasma clearance of etavopivat after a single dose | From 0 to 120 hours after investigational medicinal product (IMP) administration (day 6)
  Measured in Litre/hour (L/h).
Vz/F etavopivat: Apparent volume of distribution of etavopivat after a single dose based on plasma concentration values | From 0 to 120 hours after investigational medicinal product (IMP) administration (day 6)
  Measure in litre (L).

SECONDARY OUTCOMES:
Number of adverse events | From dosing (day 1) to end of study (day 7 to 9)
  Measured as count.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency '(dept. 2834)', Study Director — Novo Nordisk A/S
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com